CLINICAL TRIAL: NCT01268410
Title: Epidemiological Study of Patients With Acute Respiratory Failure Admitted to Brazilian Intensive Care Units
Brief Title: Epidemiology of Respiratory Insufficiency in Critical Care
Acronym: ERICC
Status: Completed | Type: Observational
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Frederico Perego Costa, Attending physincian, Hospital Sirio-Libanes
Other Study IDs: HSL2010/51
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Acute Respiratory Failure
Keywords: Acute respiratory failure; Acute lung injury; Acute respiratory distress syndrome; Mechanical Ventilation; Non-Invasive Ventilation
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute respiratory failure

SUMMARY:
Acute respiratory failure is a common entity in intensive care units nowadays and is associated with significant morbidity and mortality, thus representing a major health problem. Most of the published epidemiological studies on this condition were performed when modern ventilatory strategies and non-invasive ventilation were not available. Therefore, an actual evaluation on the incidence and outcomes of this syndrome is mandatory. We will perform an observational prospective study of patients admitted with acute respiratory insufficiency in several ICUs in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Need for non-invasive or invasive mechanical ventilation for more than 24 hours in the first 48 hours of admission to the intensive care unit.

Exclusion Criteria:

* Tracheostomized patients
* Patients admitted to ICUs for monitoring or in post-operatory of non-complicated surgeries.
* Patients with cancer on terminal stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care units in Brazil with acute respiratory failure
Sampling Method: Probability Sample
Enrollment: 773 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
hospital mortality | 15 days

SECONDARY OUTCOMES:
incidence of acute respiratory failure | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Luciano CP Azevedo, MD, PhD, Study Chair — Hospital Sirio-Libanes; Marcelo Park, MD, PhD, Principal Investigator — Hospital Sirio-Libanes; Guilherme PP Schettino, MD, PhD, Principal Investigator — Hospital Sirio-Libanes; Marcio Soares, MD, PhD, Principal Investigator — Instituto D'Or de Pesquisa e Ensino; Jorge IF Salluh, MD, PhD, Principal Investigator — Instituto D'Or de Pesquisa e Ensino
Locations (1):
- Hospital Sirio-Libanes, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Serafini SC, van Meenen DMP, Pisani L, Neto AS, Ball L, de Abreu MG, Algera AG, Azevedo L, Bellani G, Dondorp AM, Fan E, Laffey JG, Pham T, Tschernko EM, Schultz MJ, van der Woude MCE; ERICC; LUNG SAFE; PRoVENT; PRoVENT-iMiC-investigators. Different ventilation intensities among various categories of patients ventilated for reasons other than ARDS--A pooled analysis of 4 observational studies. J Crit Care. 2024 Jun;81:154531. doi: 10.1016/j.jcrc.2024.154531. Epub 2024 Feb 10. PMID 38341938
- [Derived] Azevedo LC, Park M, Salluh JI, Rea-Neto A, Souza-Dantas VC, Varaschin P, Oliveira MC, Tierno PF, dal-Pizzol F, Silva UV, Knibel M, Nassar AP Jr, Alves RA, Ferreira JC, Teixeira C, Rezende V, Martinez A, Luciano PM, Schettino G, Soares M; ERICC (Epidemiology of Respiratory Insufficiency in Critical Care) investigators. Clinical outcomes of patients requiring ventilatory support in Brazilian intensive care units: a multicenter, prospective, cohort study. Crit Care. 2013 Apr 4;17(2):R63. doi: 10.1186/cc12594. PMID 23557378